CLINICAL TRIAL: NCT06946615
Title: Exploratory Clinical Study of Combined Claudin18.2-Targeted CAR-DC and CAR-T Therapy in Patients With Advanced Colorectal Cancer
Brief Title: Exploratory Clinical Study of Claudin18.2-Targeted CAR-DC and CAR-T Therapy in Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0255
Record Dates: First submitted 2025-04-10; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Neoplasia
Keywords: Chimeric Antigen Receptor Dendritic Cells; Chimeric Antigen Receptor T-Cells; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T and CAR-DC Combination Therapy (Experimental): This arm involves the sequential administration of two biological interventions, with Claudin18.2-targeted CAR-DCs administered first, followed by Claudin18.2-targeted CAR-T cells.
  Interventions: Biological: Claudin18.2-targeted CAR-T Cells; Biological: Claudin18.2-targeted CAR-DCs

INTERVENTIONS:
Biological: Claudin18.2-targeted CAR-T Cells — Autologous T cells genetically modified to express a chimeric antigen receptor (CAR) targeting Claudin18.2.
Biological: Claudin18.2-targeted CAR-DCs — Autologous dendritic cells (DCs) genetically modified to express a chimeric antigen receptor (CAR) targeting Claudin18.2.

SUMMARY:
This is an open-label, single-arm clinical study designed to evaluate the safety and preliminary efficacy of Claudin18.2-targeted CAR-DC combined with CAR-T cell therapy in patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
Main purpose:

To evaluate the safety of Claudin18.2-targeted CAR-T cells in combination with CAR-DCs in patients with advanced colorectal cancer during the dose-escalation phase.

To determine the maximum tolerated dose of Claudin18.2-targeted CAR-DCs when administered in combination with CAR-T cells.

Secondary purpose:

To assess the overall response rate (ORR), including complete response (CR) and partial response (PR), as well as overall survival (OS) and disease-free survival (DFS) in patients receiving the combination therapy.

To evaluate the in vivo persistence, immunophenotype, and functional activity of CAR-T cells and CAR-DCs following infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a histologically or cytologically confirmed diagnosis of colonic or rectal adenocarcinoma, with at least one measurable lesion meeting RECIST v1.1 criteria (i.e., a target lesion with a longest diameter ≥10 mm on spiral CT scan, or a lymph node with a short axis ≥15 mm).
2. Claudin18.2 expression must be confirmed as positive in tumor tissue by immunohistochemistry (IHC).
3. Disease progression following standard treatments, including prior administration of fluoropyrimidines, irinotecan, and oxaliplatin. Disease progression may occur during or after treatment. Prior molecular targeted therapies are allowed.
4. ECOG performance status of 0 to 1.
5. Expected survival of at least 6 months.
6. Toxicities related to prior antitumor treatments must have resolved to baseline or ≤ Grade 1 (except for residual alopecia); peripheral neurotoxicity ≤ Grade 2 is acceptable. The minimum washout period is 4 weeks for chemotherapy and immunotherapy, and 2 weeks for targeted therapy.
7. Adequate organ function, defined as follows:

   * Hematologic function: Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelet count ≥ 75 × 10^9/L, and hemoglobin ≥ 9 g/dL. No blood transfusions, granulocyte colony-stimulating factor (G-CSF), thrombopoietin (TPO), or erythropoietin (EPO) allowed within 14 days prior to hematology testing.
   * Hepatic function: Total bilirubin (TBIL) < 1.5 × upper limit of normal (ULN); AST and ALT < 2.5 × ULN. For patients with Gilbert's syndrome, TBIL < 2 × ULN. For patients with liver metastases, AST and ALT must be < 5 × ULN.
   * Renal function: Serum creatinine ≤ 1.5 × ULN; or if > 1.5 × ULN, creatinine clearance (CrCl) ≥ 60 mL/min as calculated by the Cockcroft-Gault formula.
   * Coagulation function: Prothrombin time (PT) and activated partial thromboplastin time (APTT) < 1.5 × ULN; international normalized ratio (INR) < 1.5 or within the therapeutic range if on anticoagulation therapy.
8. Participants of childbearing potential must agree to use effective contraception during the study period.
9. Participants must have adequate comprehension and voluntarily sign the informed consent form.
10. Willingness to comply with all study-related procedures, including scheduled visits, drug administration, laboratory assessments, and other protocol requirements.

Exclusion Criteria:

1. Tumor-related emergencies requiring immediate intervention, such as malignant pericardial effusion or cardiac tamponade, superior vena cava syndrome, or spinal cord compression.
2. Clinically significant cardiovascular disease, including:

   * Documented cardiovascular events within the past 6 months, such as myocardial infarction, angina, heart failure, severe arrhythmias, or history of angioplasty, stent implantation, or coronary artery bypass grafting (CABG);
   * Prolonged QT/QTcF interval with clinical significance (QT/QTcF > 470 ms in females or > 450 ms in males).
3. Clinically significant bleeding disorders or coagulopathies, such as hemophilia.
4. Active infections including HIV, syphilis, or active hepatitis B or C:

   * Hepatitis B: HBV-DNA ≥ 1000 IU/mL;
   * Hepatitis C: Positive HCV RNA with abnormal liver function.
5. History of involuntary psychiatric hospitalization due to mental illness or other psychiatric disorders deemed unsuitable for treatment by the investigator.
6. Presence of autoimmune diseases or chronic use of immunosuppressive agents or corticosteroids.
7. Poor medication compliance or inability to adhere to the treatment protocol.
8. Any other condition that, in the opinion of the investigator, warrants exclusion from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First 3 month post CAR-T cells and CAR-DCs infusion
  To evaluate adverse events occurring within the first three months following infusion of Claudin18.2-targeted CAR-T cells and CAR-DCs. The assessment includes incidence and severity of treatment-related symptoms such as neurological toxicity, hematological abnormalities, infections, autoimmune reactions, and secondary malignancies.
Efficacy: Remission Rate | 3 months post CAR-T cells and CAR-DCs infusion
  To evaluate the proportion of participants who achieve an objective tumor response, including complete remission (CR) and partial remission (PR)

SECONDARY OUTCOMES:
Progression-Free Survival | Up to 24 months post CAR-T cells and CAR-DCs infusion
Overall Survival | Up to 24 months post CAR-T cells and CAR-DCs infusion
Relapse Rate | Up to 24 months post CAR-T cells and CAR-DCs infusion
Duration of Response | Up to 24 months post CAR-T cells and CAR-DCs infusion
In Vivo Persistence of CAR-T cells and CAR-DCs and Cytokine Profile Monitoring | First 2 weeks post CAR-T cells and CAR-DCs infusion
  The copy number of CAR-T cells and CAR-DCs in PBMCs will be measured by qPCR to assess in vivo persistence.
  Serum cytokine levels, including IL-2, IL-4, IL-6, IFN-γ, TNF-α, IL-10, IL-12, and IL-17A, will be quantified by ELISA to evaluate immune activation following cell infusion.
Objective Response Rate in Participants Receiving Different Doses of CAR-DCs | Up to 24 months post CAR-T cells and CAR-DCs infusion
  The proportion of participants in each CAR-DCs dose cohort (5×10^6, 1×10^7, 3×10^7, and 9×10^7 cells) who achieve an objective tumor response, including complete remission (CR) or partial remission (PR). All participants received a fixed dose of Claudin18.2-targeted CAR-T cells (2×10^6 cells/kg) following CAR-DCs infusion.
Incidence and Severity of Treatment-Related Adverse Events in Participants Receiving Different Doses of CAR-DCs | Up to 24 months post CAR-T cells and CAR-DCs infusion
  To evaluate adverse events occurring following infusion of Claudin18.2-targeted CAR-DCs and CAR-T cells. Participants will receive CAR-DCs at one of four dose levels (5×10^6, 1×10^7, 3×10^7, and 9×10^7 cells), followed by a fixed dose of Claudin18.2-targeted CAR-T cells (2×10^6 cells/kg). The assessment includes the incidence and severity of treatment-related symptoms such as neurological toxicity, hematological abnormalities, infections, autoimmune reactions, and secondary malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China